CLINICAL TRIAL: NCT03626467
Title: A Phase IV, Open-label, Multicenter and Single-arm on the Immunogenicity of Nonavalent Vaccine Against Human Papillomavirus in Men Infected by HIV Who Have Sex With Men. GESIDA 10017
Brief Title: A Clinical Trial to Evaluate the Immunogenicity of the Nonavalent Vaccine Against Human Papillomavirus in Men Infected by HIV Who Have Sex With Men. GESIDA 10017
Acronym: GESIDA10017
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA10017
Record Dates: First submitted 2018-07-06; First posted 2018-08-13 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: A phase IV, open-label and single-arm clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Men infected by HIV who have sex with men
  Interventions: Biological: HPV9v

INTERVENTIONS:
Biological: HPV9v — Single-arm, phase 4 study. Patients will be treated with HPV9v vaccine at baseline, week 8 and week 24
  Other Names: Gardasil9

SUMMARY:
Phase IV, open, multicenter and single-arm clinical trial designed to evaluate the immunogenicity of the HPV9v vaccine in men with HIV infection (HIV +) who have sex with men (MSM)

DETAILED DESCRIPTION:
The investigators estimate that 166 participants will need to be included in the study to evaluate the immunogenicity of vaccine against human papillomavirus in men with HIV infection who have sex with men, by evaluating in two age groups and the seroconversion rate for each of the HPV genotypes included in the vaccine from baseline to month 7 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give their written consent to participate in the study. (preferably in writing or, failing that, orally before independent witnesses of the research team) after having received information about the design, the purposes of the study, the possible risks that may arise from it and the possibility of withdrawing from it at any time. moment.
* Understand the purpose of the study and be available to perform the visits stipulated in the protocol.
* Be ≥18 years and <of 36 years.
* Patient with chronic infection with HIV-1.
* Viral HIV load <50 copies / ml and CD4> 200 cells / uL for at least the last six months.
* Transgender men or women who have had insertive or receptive anal sex with other men

Exclusion Criteria:

* Previous history of anal cancer.
* Have previously received any vaccine against HPV.

Ages: 18 Years to 36 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who serocovertize for each of the HPV genotypes included in the vaccine | From basal until week 96
  The HPV genotypes studied are: 6/11/16/18/31/33/45/52/58. The cut-off points to determine serological status 30, 16, 20, 24, 10, 8, 8, 8, and 8 units / mL for HPV genotypes 6, 11, 16, 18, 31, 33, 45, 52 , and 58, respectively

SECONDARY OUTCOMES:
Number of participants with low CD4 / CD8 ratio (<0.5) and normal ratio (> 1) | From basal until week 96
  The low CD4 / CD8 ratio has been associated with immunosenescence in the serological response, such as worse immunogenicity and worse response to vaccines
Number and type of metabolites derived from the microbiota of patients | From basal until week 96
  Detect biomarkers derived from microbiota and their relationship with the vaccine response
Percentage of participants <26 years and ≥ 26 years with persistent anal infection due to HPV | Basal, week 28 and week 96
The proportion of subjects experiencing adverse events | From basal until week 96
  Adverse events
The proportion of subjects with a severe adverse experience | From basal until week 96
  Adverse events
The proportion of subjects with an adverse experience leading to disruption | From basal until week 96
  Adverse events
The proportion of subjects with an adverse experience related to medication | From basal until week 96
  Adverse events
The proportion of subjects experiencing adverse events related to laboratory values at any time during the study period | From basal until week 96
  Adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Ramón y Cajal, Madrid
  - Hospital Fundación Jimenez Díaz, Madrid
  - Hospital La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No